CLINICAL TRIAL: NCT05398276
Title: A Tailored Exposure Intervention for Exercise Anxiety and Avoidance in Cardiac Rehabilitation
Brief Title: Behavioral Exposure for Introceptive Tolerance RCT
Acronym: BE-FIT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Samantha Farris, Ph.D., Principal Investigator, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2021000886; R01AG070136 (NIH)
Record Dates: First submitted 2022-05-26; First posted 2022-05-31 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Exercise Sensitivity; Introceptive Exposure; Anxiety; Cardiac Rehabilitation
Keywords: Exercise Sensitivity; Introceptive Exposure; Kinesiophobia; Acceptance and Commitment Therapy
MeSH Terms: conditions — Anxiety Disorders; Kinesiophobia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Exposure For Introceptive Tolerance (Experimental): The BE-FIT intervention is a cognitive-behavioral intervention and is designed to target exercise anxiety. The three main components of BE-FIT include: 1) exposure to feared bodily sensations and exercise, 2) prevention of safety behavior use before/during/after exercise, and 3) use of a wrist-worn activity monitor (Fitbit) for PA feedback and activity goal setting.
  Interventions: Behavioral: Behavioral Exposure For Introceptive Tolerance
- Health Education Control (Active Comparator): HEC is a time-matched control intervention that will be delivered on the same delivery schedule as BE-FIT. In this arm, participants will be provided educational information about health topics relevant to healthy aging delivered through PowerPoint lectures and handouts and use a Fitbit for PA monitoring.
  Interventions: Behavioral: Health Education Control

INTERVENTIONS:
Behavioral: Behavioral Exposure For Introceptive Tolerance — BE-FIT will consist of a 6-session one-on one program with a clinician that are approximately 45 minutes delivered, over the course of 3 weeks (twice/week). Sessions will coincide with scheduled cardiac rehabilitation sessions at RWJ Cardiac Rehabilitation Program. The elements of BE-FIT are (1) psychoeducation about avoidance/anxiety and values clarification and committed action for exercise and lifestyle PA; (2) graded, repeated exposure to bodily sensations and exercise to build tolerance of discomfort; (3) fading safety behaviors and elimination of exercise avoidance behaviors to promote tolerance of uncertainty and reduce catastrophizing; and (4) use of Fitbit activity tracker to facilitate physical activity monitoring and provide physical activity feedback and goal-setting.
  Other Names: BEFIT
  Arms: Behavioral Exposure For Introceptive Tolerance
Behavioral: Health Education Control — HEC is a time-matched control intervention that will be administered on the same delivery schedule as BE-FIT. The intervention content includes: (1) educational information about health topics relevant to healthy aging, and (2) Use of the Fitbit activity watch for PA monitoring. The 6 topics introduced in the HEC include: nutrition, sleep, brain health, emotional health, living with chronic conditions, how to be a smart patient. The health information will be conveyed through lectures and handouts. The goal of sessions will be to provide education, particularly as it relates to healthy aging. Patients will be given the same Fitbit as in the BE-FIT but will not be given PA goals.
  Other Names: HEC
  Arms: Health Education Control

SUMMARY:
Behavioral Exposure for Interoceptive Tolerance (BE-FIT) is a mechanism-informed behavioral intervention to target exercise anxiety. The three primary components of BE-FIT include: (1) exposure to feared bodily sensations and exercise; (2) prevention of safety behavior use before/during/after exercise, and (3) use of a wrist-worn activity monitor for physical activity (PA) feedback and activity goal setting. Evidence from the investigators' Stage I trial indicated that BE-FIT is feasible, acceptable, and safe and produced reductions in exercise anxiety and increased exercise outcomes (short-term moderate-to-vigorous intensity physical activity and steps/day). The investigators' present aim is to conduct a Stage II randomized-controlled trial to further evaluate the efficacy of BE-FIT in decreasing exercise anxiety in cardiac rehabilitation (CR) patients and examine whether changes in this target yield successive changes in exercise adherence outcomes.

DETAILED DESCRIPTION:
This study is a Stage II randomized-controlled trial of a novel behavioral intervention, titled Behavioral Exposure for Interoceptive Tolerance (BE-FIT), to evaluate (1) its efficacy in improving exercise adherence in CR and (2) its mechanisms of change in individuals 40 years of age and older. One hundred and forty-six patients enrolled in Robert Wood Johnson University Hospital (RWJ) cardiac rehabilitation (CR) program who have elevated exercise anxiety, as indicated by endorsement of much to very much concern about at least 3 items on the Exercise Sensitivity Questionnaire (ESQ; Farris et al., 2020) and meet other eligibility criteria will be randomly assigned to either receive BE-FIT, a tailored intervention specifically for CR patients with high levels of exercise anxiety (n=73), or the health education condition (HEC; n=73), which are matched for contact time. Eligible participants will be stratified based on their risk profile (determined by their electronic health record), age, sex, and ESQ score. These stratification variables were selected because they are associated with anxiety and fitness levels which could impact physical activity (PA) outcomes. Both conditions will be administered by trained doctoral-level students enrolled at Rutgers University and will be supervised throughout the course of the study by Dr. Farris and other listed co-investigators.

The BE-FIT intervention is a cognitive-behavioral intervention and is designed to target exercise anxiety. The three main components of BE-FIT include: 1) exposure to feared bodily sensations and exercise, 2) prevention of safety behavior use before/during/after exercise, and 3) use of a wrist-worn activity monitor (Fitbit) for PA feedback and activity goal setting. The alternative type of intervention is the Health Education Control (HEC), which is a time-matched control intervention that will be delivered on the same delivery schedule as BE-FIT. The doctoral-level clinicians who will be delivering HEC will be exclusively trained in order to avoid contamination with the BE-FIT intervention. In this control arm, participants will be provided educational information about health topics relevant to healthy aging delivered through PowerPoint lectures and handouts and use a Fitbit for PA monitoring. The HEC protocol has been used in prior studies conducted by Dr. Abrantes (co-investigator).

The overall duration of the study is 24 weeks, or approximately 6 months. Subjects will be involved in 6 individual sessions delivered twice weekly during the initial weeks of outpatient CR. Sessions occur for 45 minutes either immediately before or after regularly scheduled CR sessions. Five independent assessments are conducted at baseline, EOT, and three follow-ups (Weeks 12, 18, 24). Data collection will occur at each visit, with baseline data collected at the initial visit.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 40 years of age
2. Elevated exercise anxiety (score of ≥ 30 on ESQ-18)
3. Low active (< 90 min self-reported moderate-to-vigorous intensity physical activity/day in past three months)
4. Medically approved cardiac rehabilitation
5. English proficiency

Exclusion Criteria:

1. Evidence of cognitive impairment (≤ 23 on Montreal Cognitive Assessment; MoCA)
2. Severe disabling chronic medical and/or psychiatric comorbidities determined on a case-by-case basis that prevents safe or adequate participation
3. Expectation that patient will not live through study periods

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2022-05-03 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Overall minutes of exercise | 24 weeks
  Objectively measured exercise (moderate-to-vigorous intensity physical activity mins/day) on both CR and non-CR days.

SECONDARY OUTCOMES:
Percent of prescribed cardiac rehabilitation attended. | 24 weeks
Objectively measured Lifestyle PA (steps/day). | 24 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - RWJ Cardiac Rehab at East Brunswick, East Brunswick, New Jersey
  - Rutgers Emotion, Health and Behavior Laboratory Department of Psychology, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Farris SG, Kibbey MM, Derby L, Keller B, Leyro TM, Alderman BL, Steinberg MB, Abrantes AM, DiBello AM. A Confirmatory Factory Analysis of the Exercise Sensitivity Questionnaire (ESQ). J Cardiopulm Rehabil Prev. 2025 May 1;45(3):207-214. doi: 10.1097/HCR.0000000000000933. Epub 2025 Feb 28. PMID 40014001

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/76/NCT05398276/Prot_SAP_000.pdf